CLINICAL TRIAL: NCT03395197
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY OF TALAZOPARIB WITH ENZALUTAMIDE IN METASTATIC CASTRATION-RESISTANT PROSTATE CANCER
Brief Title: Talazoparib + Enzalutamide vs. Enzalutamide Monotherapy in mCRPC
Acronym: TALAPRO-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3441021; TALAPRO-2 (Other: Alias Study Number); 2023-509087-20-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2017-11-21; First posted 2018-01-10 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: mCRPC
Keywords: mCRPC (metastatic castration-resistant prostate cancer)
MeSH Terms: interventions — talazoparib; enzalutamide

STUDY DESIGN:
Intervention Model Description: To assess radiographic PFS in men with mCRPC (with no systemic treatments initiated after documentation of mCRCP) treated with talazoparib and enzalutamide vs. placebo plus enzalutamide
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination arm (Experimental): Talazoparib plus enzalutamide
  Interventions: Drug: Talazoparib with enzalutamide
- Monotherapy arm (Active Comparator): Ezalutamide plus placebo
  Interventions: Drug: Placebo with enzalutamide

INTERVENTIONS:
Drug: Talazoparib with enzalutamide — Talazoparib 0.5 mg/day plus enzalutamide 160mg/day
  Arms: Combination arm
Drug: Placebo with enzalutamide — Placebo plus enzalutamide 160 mg/day
  Arms: Monotherapy arm

SUMMARY:
This study compares rPFS in men with mCRPC treated with talazoparib plus enzalutamide vs. enzalutamide after confirmation of the starting dose of talazoparib in combination with enzalutamide.

DETAILED DESCRIPTION:
Part 1 is an open-label, non-randomized, safety and PK run-in study designed to confirm the starting dose of talazoparib in combination with enzalutamide through assessment of target safety events and PK at select sites. Part 2 is a randomized, double-blind, placebo-controlled, multinational study comparing talazoparib plus enzalutamide vs. placebo plus enzalutamide in patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed adenocarcinoma of the prostate without small cell or signet cell features

Asymptomatic or mildly symptomatic metastatic castration resistant prostate cancer (mCRPC) (score on BPI-SF Question #3 must be < 4).

For enrollment into Part 2 only (optional in Part 1): assessment of DDR mutation status

Consent to a saliva sample collection for a germline comparator unless prohibited by local regulations or ethics committee decision (optional for patients in Part 1).

Surgically or medically castrated, with serum testosterone ≤ 50 ng/dL (≤ 1.73 nmol/L) at screening.

Metastatic disease in bone documented on bone scan or in soft tissue documented on CT/MRI scan.

Progressive disease at study entry in the setting of medical or surgical castration as defined by 1 or more of the following 3 criteria:

* Prostate specific antigen (PSA) progression defined by a minimum of 2 rising PSA values from 3 consecutive assessments with an interval of at least 7 days between assessments..
* Soft tissue disease progression as defined by RECIST 1.1.
* Bone disease progression defined by Prostate Cancer Working Group 3 (PCWG3) with 2 or more new metastatic bone lesions on a whole body radionuclide bone scan.

Ongoing bisphosphonate or denosumab use prior to Day 1 (Part 1) or randomization (Part 2) is allowed but not mandatory.

Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.

Life expectancy ≥ 12 months as assessed by the investigator.

Able to swallow the study drug and have no known intolerance to study drugs or excipients.

Must agree to use a condom when having sex with a partner from the time of the first dose of study drug through 4 months after last dose of study treatment. Must also agree for female partner of childbearing potential to use an additional highly effective form of contraception from the time of the first dose of study treatment through 4 months after last dose of study treatment when having sex with a non pregnant female partner of childbearing potential.

Must agree not to donate sperm from the first dose of study drug to 4 months after the last dose of study drug.

Evidence of a personally signed and dated informed consent document (and molecular prescreening consent if appropriate) indicating that the patient [or a legally acceptable representative/legal guardian] has been informed of all pertinent aspects of the study.

Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

Any prior systemic cancer treatment initiated in in the non metastatic CRPC and mCRPC disease state.

Patients whose only evidence of metastasis is adenopathy below the aortic bifurcation.

Prior treatment with second-generation androgen receptor inhibitors (enzalutamide, apalutamide, and darolutamide), a PARP inhibitor, cyclophosphamide, or mitoxantrone for prostate cancer.

Prior treatment with platinum-based chemotherapy within 6 months (from the last dose) prior to Day 1 (Part 1) or randomization (Part 2), or any history of disease progression on platinum-based therapy within 6 months (from the last dose).

Treatment with cytotoxic chemotherapy, biologic therapy including sipuleucel T, or radionuclide therapy received in the castration-sensitive prostate cancer is NOT exclusionary if discontinued in the 28 days prior to Day 1 (Part 1) or randomization (Part 2).

Treatment with any investigational agent within 4 weeks before Day 1 (Part 1) or randomization (Part 2).

Prior treatment with opioids for pain related to either primary prostate cancer or metastasis within 28 days prior to Day 1 (Part 1) or randomization (Part 2).

Current use of potent P-gp inhibitors within 7 days prior to Day 1 (Part 1) or randomization (Part 2).

Major surgery (as defined by the investigator) within 2 weeks before Day 1 (Part 1) or randomization (Part 2), or palliative localized radiation therapy within 3 weeks before randomization (Part 2).

Clinically significant cardiovascular disease

Significant renal dysfunction as defined by any of the following laboratory abnormalities:

• Renal: eGFR < 30 mL/min/1.73 m2 by the MDRD equation (available via www.mdrd.com).

Patients enrolled in Part 1 only: Moderate renal impairment (eGFR 30-59 mL/min/1.73 m2) at screening.

Significant hepatic dysfunction as defined by any of the following laboratory abnormalities on screening labs:

* Total serum bilirubin >1.5 times the upper limit of normal (ULN) (>3 × ULN for patients with documented Gilbert syndrome or for whom indirect bilirubin concentrations suggest an extrahepatic source of elevation).
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times ULN (>5 × ULN if liver function abnormalities are due to hepatic metastasis).
* Albumin <2.8 g/dL

Absolute neutrophil count < 1500/µL, platelets < 100,000/µL, or hemoglobin < 9 g/dL (may not have received growth factors or blood transfusions within 14 days before obtaining the hematology values at screening).

Known or suspected brain metastasis or active leptomeningeal disease.

Symptomatic or impending spinal cord compression or cauda equina syndrome.

Any history of myelodysplastic syndrome, acute myeloid leukemia, or prior malignancy except any of the following:

* Carcinoma in situ or non melanoma skin cancer
* Any prior malignancies ≥3 years before randomization with no subsequent evidence of recurrence or progression regardless of the stage.
* Stage 0 or Stage 1 cancer <3 years before randomization that has a remote probability of recurrence or progression in the opinion of the investigator

Gastrointestinal disorder affecting absorption.

Fertile male subjects who are unwilling or unable to use highly effective methods of contraception for the duration of the study and for 4 months after the last dose of investigational product.

Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or patients who are Pfizer employees, including their family members, directly involved in the conduct of the study.

Other acute or chronic medical (concurrent disease, infection, or comorbidity) or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that interferes with ability to participate in the study, may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

History of seizure or any condition that may predispose to seizure (eg, prior cortical stroke, significant brain trauma). Also, history of loss of consciousness or transient ischemic attack within 12 months of randomization (Part 2).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men at least 18 years of age. For Japan, at least 20 years of age.
Enrollment: 1054 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2027-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (360):
- United States (129):
  - Alaska Urological Institute dba Alaska Clinical Research Center, Anchorage, Alaska
  - Ironwood Physicians P.C. dba Ironwood Cancer & Research Centers, Chandler, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer & Research Centers, Gilbert, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer & Research Centers, Mesa, Arizona
  - Ironwood Physicians P.C. dba Ironwood Cancer & Research Centers, Scottsdale, Arizona
  - Arizona Urology Specialists, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - South County Hematology/Oncology, Chula Vista, California
  - Sharp Rees-Stealy, Chula Vista, California
  - Glendale Adventist Medical Center, Glendale, California
  - Marin Cancer Care, Inc., Greenbrae, California
  - Cancer Center Oncology Medical Group, La Mesa, California
  - Loma Linda University Cancer Center - Records Management Only, Loma Linda, California
  - Loma Linda University Cancer Center - Hematology/Oncology Clinic, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, California
  - UCLA Clark Urology Center, Los Angeles, California
  - University of California, Irvine Medical Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - Desert Hematology Oncology Medical Group, Incorporation, Rancho Mirage, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Medical Oncology Associates-SD, San Diego, California
  - Sharp Memorial Hospital Investigational Pharmacy, San Diego, California
  - Sharp Rees-Stealy, San Diego, California
  - Stanford Health Care, Stanford, California
  - University of Colorado Denver CTO/CTRC, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Hospital- Anschutz Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital- Anschutz Outpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists, Daytona Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Lakeland Regional Health Hollis Cancer Center, Lakeland, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Lecanto, Florida
  - Florida Cancer Specialists, New Port Richey, Florida
  - Florida Cancer Specialists, Ocala, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - AdventHealth Medical Group Hermatology and Oncology, Orlando, Florida
  - Investigational Drug Services, Advent Health Orlando, Orlando, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, Spring Hill, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Stuart, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, The Villages, Florida
  - Florida Cancer Specialists, Vero Beach, Florida
  - Florida Cancer Specialists, Wellington, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Florida Cancer Specialists, Winter Park, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Piedmont Cancer Institute, Fayetteville, Georgia
  - Piedmont Cancer Institute, Newnan, Georgia
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Cook County Health (CCH), Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County/IND Pharmacy, Chicago, Illinois
  - AMITA Health Adventist Medical Center Hinsdale, Hinsdale, Illinois
  - AMITA Health Cancer Institute, Hinsdale, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Clark Memorial Hospital Radiology, Jeffersonville, Indiana
  - First Urology, PSC, Jeffersonville, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - VA Saint Louis Healthcare System, St Louis, Missouri
  - XCancer Omaha / Urology Cancer Center, PC d/b/a XCancer, Omaha, Nebraska
  - Clara Maass Medical Center, Belleville, New Jersey
  - New Jersey Cancer Care and Blood Disorders, Belleville, New Jersey
  - University Radiology, Nutley, New Jersey
  - New Jersey Urology, LLC, Voorhees Township, New Jersey
  - Urology Group of New Mexico, Albuquerque, New Mexico
  - San Juan Oncology Associates, Farmington, New Mexico
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - Montefiore Medical Center - Montefiore Medical Park, The Bronx, New York
  - TriState urologic Services PSC Inc., dba The Urology Group, Cincinnati, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Kaiser Sunnyside Medical Center, Clackamas, Oregon
  - Kaiser Westside Medical Center, Hillsboro, Oregon
  - Providence Cancer Institute Newberg Clinic, Newberg, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Cancer Institute Willamette Falls, Oregon City, Oregon
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic - Westside, Portland, Oregon
  - Providence St Vincent Medical Center - Investigational Drug Service, Portland, Oregon
  - Providence St Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - UPMC Hillman Cancer Center - Altoona, Altoona, Pennsylvania
  - UPMC Hillman Cancer Center - Upper St. Clair, Bethel Park, Pennsylvania
  - UPMC Hillman Cancer Center - Arnold Palmer - Mt View, Greensburg, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant (HOA), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant (OHA), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center - Northwest, Seneca, Pennsylvania
  - UPMC Hillman Cancer Center - Uniontown, Uniontown, Pennsylvania
  - UPMC Hillman Cancer Center - Washington, Washington, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Tennessee Oncology PLLC - Greco-Hainesworth Centers for Research, Chattanooga, Tennessee
  - Urology Associates P.C., Nashville, Tennessee
  - The Vanderbilt Clinic, Nashville, Tennessee
  - Vanderbuilt University Medical Center, Department of Urology, Nashville, Tennessee
  - Urology Austin PLLC, Austin, Texas
  - Rio Grande Urology, P.A., El Paso, Texas
  - Houston Metro Urology, Houston, Texas
  - Urology Austin, PLLC, Round Rock, Texas
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
  - Farmington Health Center -University of Utah, Farmington, Utah
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Redwood Health Center-University of Utah, Salt Lake City, Utah
  - South Jordan Health Center -University of Utah, South Jordan, Utah
  - Inova Schar Cancer Institute Infusion Pharmacy, Fairfax, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
- Argentina (6):
  - Centro de Investigacion Pergamino SA - Clinica Pergamino SA, Pergamino, Buenos Aires
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Hospital Británico de Buenos Aires, Caba
  - Centro de Educacion Medica e Investigaciones Clinicas "Norberto Quirno" Cemic, Caba
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
- Australia (13):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - River City Pharmacy, Auchenflower, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - ICON Cancer Centre Chermside, Chermside, Queensland
  - ICON Cancer Centre South Brisbane, South Brisbane, Queensland
  - Integrated Clinical Oncology Network Pty Ltd (ICON), South Brisbane, Queensland
  - ICON Cancer Centre Southport, Southport, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, North Melbourne, Victoria
- Belgium (6):
  - AZ Klina, Brasschaat
  - A.Z. Sint-Lucas, Ghent
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - Clinique Saint-Pierre Ottignies, Ottignies
  - CHU UCL Namur site Godinne, Yvoir
- Brazil (18):
  - Instituto Nacional de Câncer José de Alencar Gomes da Silva - INCA, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitario Pedro Ernesto-Centro de Pesquisas (CEPUSA), Rio de Janeiro, Rio de Janeiro
  - Hospital CopaDor, Rio de Janeiro, Rio de Janeiro
  - Hospital Gloria D'Or, Rio de Janeiro, Rio de Janeiro
  - Oncologia D'Or, Rio de Janeiro, Rio de Janeiro
  - Instituto D'Or de Pesquisa e Ensino, Rio de Janeiro, Rio de Janeiro
  - Associacao Hospital de Caridade de Ijui, Ijuí, Rio Grande do Sul
  - Sociedade Beneficencia e Caridade de Lajeado - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Centro de Pesquisa Clinica em Oncologia - Hospital Sao Lucas da Pontificia Universidade Catolica, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - MedPlex Eixo Norte, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao - Grupo Hospitalar Conceicao, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Faculdade de Medicina do ABC - Centro de Estudos e Pesquisa de Hematologia e Oncologia (CEPHO), Santo André, São Paulo
  - Faculdade de Medicina do ABC - Centro de Estudos e Pesquisas de Hematologia e Oncologia (CEPHO), Santo André, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Alemão Oswaldo Cruz, São Paulo, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo-ICESP-Nucleo de Pesquisa, São Paulo, SÃO Paulo (SP)
- Canada (8):
  - Arthur J.E Child Comprehensive Cancer Centre, Calgary, Alberta
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Centre integre universitaire de sante et de services sociaux du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre intégré universitaire de santé et de services sociaux du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Centre integre universitaire de sante et de services sociaux de l'Estrie, Sherbrooke, Quebec
- Chile (4):
  - Centro de Investigacion Clinica del Sur, Temuco, Región de la Araucanía
  - Centro de Investigaciones Clinicas Vina del Mar, Viña del Mar, Región de Valparaíso
  - Sociedad Prosalud Montes y Orlandi Ltda. Fantasy name (Orlandi Oncologia), Santiago, Santiago Metropolitan
  - James Lind Centro de Investigación del Cáncer, Araucania
- China (34):
  - The First affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou, Fujian
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Union Hospital, Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital , The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The first affiliated hospital of Ningbo university, Ningbo, Zhejiang
  - Urinary surgery, Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Hospital, Beijing
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University First Hospital / Urology Department, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Fudan University Cancer Hospital, Deptartment of Urology, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - The Fifth People's Hospital of Shanghai, Fudan University, Shanghai
  - The Second Hospital of Tianjin Medical University, Tianjin
- Czechia (4):
  - Fakultní nemocnice Hradec Králové, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Multiscan s.r.o., Pardubice
  - Fakultní nemocnice Královské Vinohrady, Prague
- Finland (7):
  - HUS Helsinki University Hospital, Helsinki
  - Docrates Cancer Center, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulun yliopistollinen sairaala, Oulu
  - Pirkanmaan hyvinvointialue, Tampere
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (14):
  - Clinique Victor Hugo Le Mans, Le Mans, Pays de la Loire Region
  - Centre d'Oncologie du Pays-Basque, Bayonne
  - Clinique Ramsay Belharra, Bayonne
  - Hopital Saint Andre - CHU de Bordeaux, Bordeaux
  - CHD Vendée, La Roche-sur-Yon
  - Centre Leon Berard, Lyon
  - Centre Léon Bérard, Lyon
  - CHU Montpellier-Hopital Saint Eloi, Montpellier
  - Hopital Saint-Louis, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Clinique Sainte Anne, Strasbourg
  - Hopitaux Universitaires de Strasbourg - ICANS, Strasbourg
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinik Heidelberg, Heidelberg
  - Universitatsklinikum Heidelberg, Heidelberg
  - Diagnostikzentrum, Kirchheim
  - Universitaetsklinikum Muenster, Münster
  - Studienpraxis Urologie, Nürtingen
- Hungary (6):
  - Semmelweis Egyetem Urologiai Klinika, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Uzsoki Utcai Korhaz, Budapest
  - Uzsoki Utcai Kórház, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont Onkoterapias Intezet, Pécs
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Azienda Ospedaliero-Universitaria Policlinico Sant' Orsola Malpighi, Bologna, BO
  - ASST di Cremona, Cremona, CR
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola, FC
  - Azienda Ospedaliera S. Maria, Terni, TN
  - Ospedale Santa Chiara, Trento, TN
  - AOU San Luigi Gonzaga, Orbassano, TO
  - Azienda Provinciale per i Servizi Sanitari, della Provincia Autonoma di Trento, Trento, Trentino-Alto Adige
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale - Napoli, Napoli
- Japan (23):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hirosaki University School of Medicine & Hospital, Hirosaki, Aomori
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kure Medical Center and Chugoku Cancer Center, Kure, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kagoshima University Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Tokushima University Hospital, Tokushima
  - Yamagata Prefectural Central Hospital, Yamagata
  - Yamagata University Hospital, Yamagata
- New Zealand (4):
  - Tauranga Urology Research Limited, Tauranga, Bay of Plenty
  - Canterbury District Health Board, Christchurch, Canterbury
  - Waikato Hospital, Hamilton, Waikato Region
  - Auckland City Hospital, Auckland
- Norway (6):
  - Sykehusapoteket Ostfold, Kalnes, Grålum
  - Ostfold County Hospital, Kalnes, Grålum
  - Akershus University Hospital, Lorenskog
  - Oslo University Hospital -Ullevål & Radiumhospitalet, Oslo
  - St. Olavs Hospital, Trondheim University Hospital, Trondheim
  - Trondheim Hospital Pharmacy, Trondheim
- Peru (4):
  - Clinica Monte Carmelo S.C.R.LTDA., Arequipa
  - Hospital Militar Central "Coronel Luis Arias Schreiber", Lima
  - Clinica Internacional Sede San Borja, Lima
  - Clinica Oncosalud, Lima
- Poland (6):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im. ks. B. Markiewicza, Brzozów
  - Szpitale Pomorskie Sp. z o.o. Oddzial Onkologii i Radioterapii, Gdynia
  - Przychodnia Lekarska "Komed" Roman Karaszewski, Konin
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Otwock
  - City Clinic Sp. z o.o., Warsaw
  - NZOZ Szpital Mazovia; Oddzial urologiczny, Warsaw
- Portugal (6):
  - Centro Clínico Académico - Braga, Associação (2CABraga), Braga
  - Instituto Português Oncologia de Coimbra Francisco Gentil - E.P.E, Coimbra
  - Fundação Champalimaud, Lisbon
  - Hospital da Luz Lisboa, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo Antonio, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, Porto
- South Africa (6):
  - Cancercare Langenhoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - The Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Wits Clinical Research, Parktown, Gauteng
  - Cancercare Rondebosch Oncology, Cape Town, Western Cape
  - Outeniqua Cancercare Oncology Unit, George, Western Cape
  - Cape Town Oncology Trials, Kraaifontein, Western Cape
- South Korea (13):
  - Clinical Trial Pharmacy, National Cancer Center, Goyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Clinical Trial Center, Serverance Hospital, yonsei University Health System, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Cancer Center Clinical Trial, Asan Medical Center, Seoul
  - Clinical Trials Center Pharmacy, Seoul
  - Samsung Medical Center, Seoul
  - Clinical Trial Pharmacy, The Catholic University of Korea, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (11):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital General Universitario de Elche, Elche, Alicante
  - Institut Catala d'Oncologia - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Corporacio Sanitaria i Universitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario 12 De Octubre, Madrid
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands LÄN [se-14]
  - Karolinska Universitetssjukhuset, Solna
  - Cancercentrum, Umeå
- United Kingdom (11):
  - University Hospitals Plymouth NHS Trust, Plymouth, Devon
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - Greater Glasgow Health Board J B Russell House, Gartnavel Royal Hospital, Glasgow, Scotland
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - Royal Cornwall Hospitals NHS Trust, Cornwall
  - NHS Greater Glasgow and Clyde (Radiology/Scans Address), Glasgow
  - NHS Greater Glasgow and Clyde, The Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre - Liverpool, Liverpool
  - Imperial College Healthcare NHS Trust, London
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, London
  - Department of Oncology, Cancer and Haematology Centre, Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Agarwal N, Azad AA, Carles J, Fay AP, Matsubara N, Szczylik C, De Giorgi U, Young Joung J, Fong PCC, Voog E, Jones RJ, Shore ND, Saad F, Dunshee C, Zschabitz S, Oldenburg J, Lin X, Healy CG, Kalac M, Kennedy D, Fizazi K. Talazoparib plus enzalutamide in men with metastatic castration-resistant prostate cancer: final overall survival results from the randomised, placebo-controlled, phase 3 TALAPRO-2 trial. Lancet. 2025 Aug 2;406(10502):447-460. doi: 10.1016/S0140-6736(25)00684-1. Epub 2025 Jul 16. PMID 40683290
- [Derived] Fizazi K, Azad AA, Matsubara N, Carles J, Fay AP, De Giorgi U, Young Joung J, Fong PCC, Voog E, Jones RJ, Shore ND, Dunshee C, Zschabitz S, Oldenburg J, Ye D, Lin X, Kalac M, Douglas Laird A, Kennedy D, Agarwal N. Talazoparib plus enzalutamide in men with HRR-deficient metastatic castration-resistant prostate cancer: final overall survival results from the randomised, placebo-controlled, phase 3 TALAPRO-2 trial. Lancet. 2025 Aug 2;406(10502):461-474. doi: 10.1016/S0140-6736(25)00683-X. Epub 2025 Jul 16. PMID 40683287
- [Derived] Fay AP, Fizazi K, Matsubara N, Azad AA, Saad F, De Giorgi U, Joung JY, Fong PCC, Jones RJ, Zschabitz S, Oldenburg J, Shore ND, Dunshee C, Carles J, Cislo P, Chang J, Healy CG, Niyazov A, Agarwal N. First-line talazoparib plus enzalutamide versus placebo plus enzalutamide in men with metastatic castration-resistant prostate cancer and homologous recombination repair gene alterations: patient-reported outcomes from the randomised, double-blind, placebo-controlled, phase 3 TALAPRO-2 trial. Lancet Oncol. 2025 Apr;26(4):481-490. doi: 10.1016/S1470-2045(25)00031-2. PMID 40179907
- [Derived] Matsubara N, Azad AA, Agarwal N, Saad F, De Giorgi U, Joung JY, Fong PCC, Jones RJ, Zschabitz S, Oldenburg J, Shore ND, Dunshee C, Carles J, Fay AP, Cislo P, Chang J, Healy CG, Niyazov A, Fizazi K. First-line talazoparib plus enzalutamide versus placebo plus enzalutamide for metastatic castration-resistant prostate cancer: patient-reported outcomes from the randomised, double-blind, placebo-controlled, phase 3 TALAPRO-2 trial. Lancet Oncol. 2025 Apr;26(4):470-480. doi: 10.1016/S1470-2045(25)00030-0. PMID 40179906
- [Derived] Matsubara N, Miyake H, Uemura H, Mizokami A, Kikukawa H, Kosaka T, Nishimura K, Nakamura M, Kobayashi K, Komaru A, Mori Y, Toyoizumi S, Hori N, Umeyama Y, Uemura H. Phase 3 Study of Talazoparib Plus Enzalutamide Versus Placebo Plus Enzalutamide as First-Line Treatment in Patients With Metastatic Castration-Resistant Prostate Cancer: TALAPRO-2 Japanese Subgroup Analysis. Cancer Med. 2025 Jan;14(1):e70333. doi: 10.1002/cam4.70333. PMID 39737542
- [Derived] Azad AA, Fizazi K, Matsubara N, Saad F, De Giorgi U, Joung JY, Fong PCC, Jones RJ, Zschabitz S, Oldenburg J, Shore ND, Dunshee C, Carles J, Fay AP, Lin X, DeAnnuntis L, Di Santo N, Zielinski MA, Agarwal N. Talazoparib plus enzalutamide in metastatic castration-resistant prostate cancer: Safety analyses from the randomized, placebo-controlled, phase III TALAPRO-2 study. Eur J Cancer. 2024 Dec;213:115078. doi: 10.1016/j.ejca.2024.115078. Epub 2024 Oct 20. PMID 39486165
- [Derived] Agarwal N, Saad F, Azad AA, Mateo J, Matsubara N, Shore ND, Chakrabarti J, Chen HC, Lanzalone S, Niyazov A, Fizazi K. The TALAPRO-3 study design: a plain language summary. Future Oncol. 2024;20(30):2225-2231. doi: 10.1080/14796694.2024.2363131. Epub 2024 Jul 24. PMID 39451095
- [Derived] Agarwal N, Azad AA, Carles J, Fay AP, Matsubara N, Heinrich D, Szczylik C, De Giorgi U, Joung JY, Fong PCC, Voog E, Jones RJ, Shore ND, Dunshee C, Zschabitz S, Oldenburg J, Lin X, Healy CG, Di Santo N, Zohren F, Fizazi K. Plain language summary of the results from the TALAPRO-2 study: Talazoparib plus enzalutamide versus placebo plus enzalutamide for patients with advanced prostate cancer. Future Oncol. 2024;20(29):2123-2135. doi: 10.1080/14796694.2024.2362108. Epub 2024 Jul 12. PMID 38995237
- [Derived] Heiss BL, Chang E, Gao X, Truong T, Brave MH, Bloomquist E, Shah A, Hamed S, Kraft J, Chiu HJ, Ricks TK, Tilley A, Pierce WF, Tang L, Abukhdeir A, Kalavar S, Philip R, Tang S, Pazdur R, Amiri-Kordestani L, Kluetz PG, Suzman DL. US Food and Drug Administration Approval Summary: Talazoparib in Combination With Enzalutamide for Treatment of Patients With Homologous Recombination Repair Gene-Mutated Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2024 May 20;42(15):1851-1860. doi: 10.1200/JCO.23.02182. Epub 2024 Mar 7. PMID 38452327
- [Derived] Fizazi K, Azad AA, Matsubara N, Carles J, Fay AP, De Giorgi U, Joung JY, Fong PCC, Voog E, Jones RJ, Shore ND, Dunshee C, Zschabitz S, Oldenburg J, Ye D, Lin X, Healy CG, Di Santo N, Laird AD, Zohren F, Agarwal N. First-line talazoparib with enzalutamide in HRR-deficient metastatic castration-resistant prostate cancer: the phase 3 TALAPRO-2 trial. Nat Med. 2024 Jan;30(1):257-264. doi: 10.1038/s41591-023-02704-x. Epub 2023 Dec 4. PMID 38049622
- [Derived] Agarwal N, Azad AA, Carles J, Fay AP, Matsubara N, Heinrich D, Szczylik C, De Giorgi U, Young Joung J, Fong PCC, Voog E, Jones RJ, Shore ND, Dunshee C, Zschabitz S, Oldenburg J, Lin X, Healy CG, Di Santo N, Zohren F, Fizazi K. Talazoparib plus enzalutamide in men with first-line metastatic castration-resistant prostate cancer (TALAPRO-2): a randomised, placebo-controlled, phase 3 trial. Lancet. 2023 Jul 22;402(10398):291-303. doi: 10.1016/S0140-6736(23)01055-3. Epub 2023 Jun 4. PMID 37285865
- [Derived] Agarwal N, Azad A, Shore ND, Carles J, Fay AP, Dunshee C, Karsh LI, Paccagnella ML, Santo ND, Elmeliegy M, Lin X, Czibere A, Fizazi K. Talazoparib plus enzalutamide in metastatic castration-resistant prostate cancer: TALAPRO-2 phase III study design. Future Oncol. 2022 Feb;18(4):425-436. doi: 10.2217/fon-2021-0811. Epub 2022 Jan 26. PMID 35080190
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: As of the data cutoff for the primary completion date (PCD) on 16 Aug 2022 for Part 1 and Part 2 Cohort 1 and on 03 Oct 2022 for Part 2 Cohort 2, for overall study, 2896 participants were screened for participation in the C3441021 study. As of 03 Oct 2022, a total of 1054 participants were enrolled in this study.
Pre-assignment Details: As of 16 Aug 2022, 19 participants were enrolled in Part 1, 805 participants with metastatic castrate-resistant prostate cancer (mCRPC) unselected for DNA damage response (DDR) deficiencies were randomized in Part 2 Cohort 1. As of 03 Oct 2022, 169 DDR-deficient participants enrolled in Cohort 1 were combined with the 230 DDR-deficient participants enrolled in Cohort 2 such that 399 participants were included in the analysis for participants with DDR deficiencies.
Groups:
- Part 1: Talazoparib 1 mg QD+Enzalutamide: Participants initially received a starting dose of talazoparib 1 mg once daily (QD) in combination with enzalutamide 160 mg QD up until Day 66, then the dose of talazoparib was reduced to 0.5 mg QD based on results from a review of available safety and pharmacokinetic (PK) data (up to a maximum of 231.14 weeks for both talazoparib and enzalutamide as of 16 Aug 2022).
- Part 1: Talazoparib 0.5 mg QD+Enzalutamide: Participants received talazoparib 0.5 mg QD in combination with enzalutamide 160 mg QD (up to a maximum of 180 weeks for talazoparib and 219.29 weeks for enzalutamide as of 16 Aug 2022).
- Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer): Participants were randomized to receive talazoparib 0.5 mg QD in combination with enzalutamide 160 mg QD (up to a maximum of 186.14 weeks for both talazoparib and enzalutamide as of 16 Aug 2022).
- Part 2 Cohort 1: Placebo+Enzalutamide (All-comer): Participants were randomized to receive placebo QD in combination with enzalutamide 160 mg QD (up to a maximum of 182 weeks for both placebo and enzalutamide as of 16 Aug 2022).
- Part 2 Cohort 2: Talazoparib+Enzalutamide (DDR-deficient): Participants with DDR deficiencies were randomized to receive talazoparib 0.5 mg QD in combination with enzalutamide 160 mg QD (up to a maximum of 169.86 weeks for both talazoparib and enzalutamide as of 03 Oct 2022).
- Part 2 Cohort 2: Placebo+Enzalutamide (DDR-deficient): Participants with DDR deficiencies were randomized to receive placebo QD in combination with enzalutamide 160 mg QD (up to a maximum of 157 weeks for both placebo and enzalutamide as of 03 Oct 2022).
Period: Study Recruitment
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide | Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer) | Part 2 Cohort 1: Placebo+Enzalutamide (All-comer) | Part 2 Cohort 2: Talazoparib+Enzalutamide (DDR-deficient) | Part 2 Cohort 2: Placebo+Enzalutamide (DDR-deficient)
Started | 13 | 6 | 402 | 403 | 115 | 115
Completed | 13 | 6 | 402 | 403 | 115 | 115
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Analysis for Part 1 and Part 2 Cohort 1
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide | Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer) | Part 2 Cohort 1: Placebo+Enzalutamide (All-comer) | Part 2 Cohort 2: Talazoparib+Enzalutamide (DDR-deficient) | Part 2 Cohort 2: Placebo+Enzalutamide (DDR-deficient)
Started | 13 | 6 | 402 | 403 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 13 | 6 | 402 | 403 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 8 | 10 | 0 | 0
Not completed — No longer meets eligibility ceriteria | 0 | 0 | 1 | 0 | 0 | 0
Not completed — No longer clinically benefiting | 0 | 0 | 14 | 21 | 0 | 0
Not completed — Not treated with talazoparib | 0 | 0 | 5 | 3 | 0 | 0
Not completed — Adverse Event | 9 | 3 | 69 | 43 | 0 | 0
Not completed — Progressive Disease | 1 | 1 | 76 | 124 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 29 | 30 | 0 | 0
Not completed — Global Deterioration Of Health Status | 1 | 0 | 44 | 46 | 0 | 0
Not completed — Other | 1 | 1 | 4 | 5 | 0 | 0
Not completed — Ongoing | 1 | 0 | 152 | 120 | 0 | 0
Period: Analysis for DDR-Deficient Participants
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide | Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer) | Part 2 Cohort 1: Placebo+Enzalutamide (All-comer) | Part 2 Cohort 2: Talazoparib+Enzalutamide (DDR-deficient) | Part 2 Cohort 2: Placebo+Enzalutamide (DDR-deficient)
Started | 0 | 0 | 0 | 0 | 200 (Participants who were DDR-deficient and received talazoparib+enzalutamide in Part 2 Cohort 1 (85 total) were combined with participants enrolled in Part 2 Cohort 2 (115 total) and included in the analysis of discontinuation reasons for participants with DDR deficiencies (combined 200 total).) | 199 (Participants who were DDR-deficient and received placebo+enzalutamide in Part 2 Cohort 1 (84 total) were combined with participants enrolled in Part 2 Cohort 2 (115 total) and included in the analysis of discontinuation reasons for participants with DDR deficiencies (combined 199 total).)
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 200 | 199
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 4
Not completed — No longer clinically benefiting | 0 | 0 | 0 | 0 | 5 | 8
Not completed — Not treated with talazoparib | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 19 | 11
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 39 | 60
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 11 | 13
Not completed — Global Deterioration Of Health Status | 0 | 0 | 0 | 0 | 24 | 40
Not completed — Other | 0 | 0 | 0 | 0 | 3 | 3
Not completed — Ongoing | 0 | 0 | 0 | 0 | 95 | 60

BASELINE CHARACTERISTICS:
Population: Included all participants who received at least 1 dose of study treatment (talazoparib or enzalutamide) in Part 1, and all participants who were randomized to double-blind study treatment in Part 2 regardless of whether or not treatment was administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide | Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer) | Part 2 Cohort 1: Placebo+Enzalutamide (All-comer) | Part 2 Cohort 2: Talazoparib+Enzalutamide (DDR-deficient) | Part 2 Cohort 2: Placebo+Enzalutamide (DDR-deficient) | Total
Number analyzed (Participants) | 13 | 6 | 402 | 403 | 115 | 115 | 1054
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 1 | 2 | 79 | 94 | 25 | 26 | 227
  65-<75 years | 8 | 4 | 188 | 175 | 53 | 55 | 483
  >=75 years | 4 | 0 | 135 | 134 | 37 | 34 | 344
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 13 | 6 | 402 | 403 | 115 | 115 | 1054
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 6 | 243 | 255 | 88 | 90 | 694
  Black or African American | 0 | 0 | 11 | 5 | 4 | 3 | 23
  Asian | 0 | 0 | 127 | 120 | 13 | 12 | 272
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 1 | 1 | 0 | 4
  Not Reported | 0 | 0 | 19 | 21 | 8 | 10 | 58
  Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Multiracial | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Occuring Within the First 66 Days of Dosing - Part 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. TEAEs are defined as newly occurring AEs or those worsening after first dose. As per Common Terminology Criteria for Adverse Events (CTCAE) version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE. Serious TEAE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. SAEs were determined according to the investigator's assessment. Results as of 16 Aug 2022 are reported.
Time Frame: Post dose on Day 1 up to Day 66 in Part 1
Population: Included all participants in Part 1 who received at least 1 dose of study intervention (talazoparib or enzalutamide).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide
Number analyzed (Participants) | 13 | 6
Participants
  Participants with TEAEs | 13 | 6
  Participants with medication error TEAE | 0 | 0
  Participants with serious TEAE | 1 | 0
  Participants with Maximum Grade 3 or 4 TEAE | 8 | 1
  Participants with Maximum Grade 5 TEAE | 0 | 0

2. Primary Outcome: Number of Participants With All-Causality Clustered Treatment-Emergent Cytopenias by Preferred Term (PT) and Max CTCAE Grade Occuring Within the First 66 Days of Dosing - Part 1
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. TEAEs are defined as newly occurring AEs or those worsening after first dose. As per CTCAE version 4, Grade 1=mild AE; Grade 2=moderate AE; Grade 3=severe AE; Grade 4=life-threatening or disabling AE; Grade 5=death related to an AE. Medical Dictionary for Regulatory Activities (MedDRA) v25.0 coding dictionary applied. PTs for the cluster terms are: ANEMIA, including Anemia, Hematocrit decreased, Hemoglobin decreased, and Red blood cell count decreased; THROMBOCYTOPENIA, including, Thrombocytopenia and Platelet count decreased; NEUTROPENIA, including Febrile neutropenia, Neutropenia and Neutrophil count decreased; LEUKOPENIA, including Leukopenia, White blood cell count decreased. Events in any grade with at least 1 occurrence in participants are reported for this outcome measure. Results as of 16 Aug 2022 are reported.
Time Frame: Post dose on Day 1 up to Day 66 in Part 1
Population: Included all participants in Part 1 who received at least 1 dose of study intervention (talazoparib or enzalutamide).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide
Number analyzed (Participants) | 13 | 6
Participants
  Grade 2 Anemia | 2 | 0
  Grade 3 Anemia | 6 | 1
  Grade 1 Neutropenia | 1 | 0
  Grade 2 Neutropenia | 1 | 0
  Grade 3 Neutropenia | 4 | 0
  Grade 2 Leukopenia | 1 | 0
  Grade 3 Leukopenia | 3 | 0
  Grade 3 Thrombocytopenia | 2 | 0

3. Primary Outcome: Number of Participants With All-Causality TEAEs During the Overall Period of Part 1
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. TEAEs are defined as newly occurring AEs or those worsening after first dose. As per CTCAE version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE. Serious TEAE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. SAEs were determined according to the investigator's assessment. Results as of 16 Aug 2022 are reported.
Time Frame: Post dose on Day 1 up to 28 days after the last dose of study intervention, or before new systemic antineoplastic therapy, whichever occurred first (maximum of 235.14 weeks)
Population: Included all participants in Part 1 who received at least 1 dose of study intervention (talazoparib or enzalutamide).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide
Number analyzed (Participants) | 13 | 6
Participants
  Participants with TEAEs | 13 | 6
  Participants with medication error TEAE | 0 | 0
  Participants with serious TEAE | 6 | 3
  Participants with Maximum Grade 3 or 4 TEAE | 11 | 6
  Participants with Maximum Grade 5 TEAE | 1 | 0

4. Primary Outcome: Number of Participants With Treatment-Related TEAEs During the Overall Period of Part 1
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. TEAEs are defined as newly occurring AEs or those worsening after first dose. Treatment-related AE was any untoward medical occurrence attributed to study intervention in a participant who received study intervention. As per CTCAE version 4, Grade 1= mild AE; Grade 2= moderate AE; Grade 3= severe AE; Grade 4= life-threatening or disabling AE; Grade 5= death related to an AE. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. SAEs were determined according to the investigator's assessment. Results as of 16 Aug 2022 are reported.
Time Frame: as for outcome 3
Population: Included all participants in Part 1 who received at least 1 dose of study intervention (talazoparib or enzalutamide).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide
Number analyzed (Participants) | 13 | 6
Participants
  Participants with TEAEs | 13 | 6
  Participants with medication error TEAE | 0 | 0
  Participants with serious TEAE | 2 | 1
  Participants with Maximum Grade 3 or 4 TEAE | 10 | 4
  Participants with Maximum Grade 5 TEAE | 1 | 0

5. Primary Outcome: Number of Participants With All-Causality Clustered Treatment-Emergent Cytopenias by PT and Max CTCAE Grade Occuring Anytime After Dosing - Part 1
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. TEAEs are defined as newly occurring AEs or those worsening after first dose. As per CTCAE version 4, Grade 1=mild AE; Grade 2=moderate AE; Grade 3=severe AE; Grade 4=life-threatening or disabling AE; Grade 5=death related to an AE. MedDRA v25.0 coding dictionary applied. PTs for the cluster terms are: ANEMIA, including Anemia, Hematocrit decreased, Hemoglobin decreased, and Red blood cell count decreased; THROMBOCYTOPENIA, including, Thrombocytopenia and Platelet count decreased; NEUTROPENIA, including Febrile neutropenia, Neutropenia and Neutrophil count decreased; LEUKOPENIA, including Leukopenia, White blood cell count decreased. Events in any grade with at least 1 occurrence in participants are reported for this outcome measure. Results as of 16 Aug 2022 are reported.
Time Frame: as for outcome 3
Population: Included all participants in Part 1 who received at least 1 dose of study intervention (talazoparib or enzalutamide).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide
Number analyzed (Participants) | 13 | 6
Participants
  Grade 3 Anemia | 10 | 3
  Grade 1 Neutropenia | 1 | 0
  Grade 2 Neutropenia | 1 | 0
  Grade 3 Neutropenia | 6 | 0
  Grade 2 Leukopenia | 1 | 0
  Grade 3 Leukopenia | 5 | 0
  Grade 3 Thrombocytopenia | 3 | 0
  Grade 4 Anemia | 0 | 1
  Grade 2 Lymphopenia | 1 | 0
  Grade 3 Lymphopenia | 2 | 0

6. Primary Outcome: Number of Participants With Treatment-Related Clustered Treatment-Emergent Cytopenias by PT and Max CTCAE Grade in >=10% of Participants Occuring Anytime After Dosing - Part 1
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. TEAEs are newly occurring AEs or those worsening after first dose. Treatment-related AE was any AE attributed to study intervention in a participant who received study intervention. As per CTCAE version 4, Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling; Grade 5=death related to an AE. MedDRA v25.0 coding dictionary applied. PTs for the cluster terms are: ANEMIA, including Anemia, Hematocrit decreased, Hemoglobin decreased, and Red blood cell count decreased; THROMBOCYTOPENIA, including, Thrombocytopenia and Platelet count decreased; NEUTROPENIA, including Febrile neutropenia, Neutropenia and Neutrophil count decreased; LEUKOPENIA, including Leukopenia, White blood cell count decreased. Events in any grade with incidence in >=10% of participants are reported. Results as of 16 Aug 2022 are reported.
Time Frame: as for outcome 3
Population: Included all participants in Part 1 who received at least 1 dose of study intervention (talazoparib or enzalutamide).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide
Number analyzed (Participants) | 13 | 6
Participants
  Grade 3 Anemia | 10 | 3
  Grade 1 Neutropenia | 1 | 0
  Grade 2 Neutropenia | 1 | 0
  Grade 3 Neutropenia | 6 | 0
  Grade 2 Leukopenia | 2 | 0
  Grade 3 Leukopenia | 4 | 0
  Grade 3 Thrombocytopenia | 3 | 0
  Grade 4 Anemia | 0 | 1
  Grade 2 Lymphopenia | 1 | 0
  Grade 3 Lymphopenia | 2 | 0

7. Primary Outcome: Blinded Independent Central Review (BICR) Assessed Radiographic Progression-Free Survival (rPFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for All-Comers - Part 2 Cohort 1
Description: rPFS is defined as the time from the date of randomization to first objective evidence of radiographic progression as assessed in soft tissue per RECIST 1.1, or death, whichever occurs first. Soft tissue disease status was assessed at regular intervals during the course of the study by computed tomography (CT) of chest and CT or magnetic resonance imaging (MRI) of abdomen and pelvis. Progression is defined using RECIST 1.1 as a >=20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Results as of 16 Aug 2022 are reported for this outcome measure.
Time Frame: From the start of treatment to the time of first documented progression, or death (maximum up to 42 months)
Population: Included all participants randomized to double-blind study treatment in Part 2 Cohort 1 regardless of whether or not treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part 2 Cohort 1: Talazoparib+Enzalutamide: Participants were randomized to receive talazoparib 0.5 mg QD in combination with enzalutamide 160 mg QD (up to a maximum of 186.14 weeks for both talazoparib and enzalutamide as of 16 Aug 2022).
- Part 2 Cohort 1: Placebo+Enzalutamide: Participants were randomized to receive placebo QD in combination with enzalutamide 160 mg QD (up to a maximum of 182 weeks for both placebo and enzalutamide as of 16 Aug 2022).
Arm/Group | Part 2 Cohort 1: Talazoparib+Enzalutamide | Part 2 Cohort 1: Placebo+Enzalutamide
Number analyzed (Participants) | 402 | 403
Months | NA [27.5 to NA] — NA indicates not estimated due to less than half of participants meeting the criterion as of data cutoff date (16 Aug 2022). | 21.9 [16.6 to 25.1]
Statistical Analysis 1: Comparison: Part 2 Cohort 1: Talazoparib+Enzalutamide vs Part 2 Cohort 1: Placebo+Enzalutamide; The following statistical hypotheses was tested to address the primary objectives: H01: HRrPFS ≥1 vs H11: HRrPFS <1, where HRrPFS and HRrPFS+ are the hazard ratios (talazoparib in combination with enzalutamide vs. placebo in combination with enzalutamide) of rPFS based on BICR assessment in the all-comers population for Part 2 Cohort 1; Test type: Superiority; p < 0.0001, Log Rank — 1-sided; Hazard Ratio (HR) = 0.627, 95% CI 2-sided [0.506 to 0.777] — Hazard ratio was based on Cox proportional hazards model; under proportional hazards, if hazard ratio < 1, it indicates reduction in hazard rate in favor of Talazoparib+Enzalutamide compared to Placebo+Enzalutamide

8. Primary Outcome: BICR Assessed rPFS Per RECIST 1.1 in Patients With DDR Deficiencies - Part 2
Description: rPFS is defined as the time from the date of randomization to first objective evidence of radiographic progression as assessed in soft tissue per RECIST 1.1, or death, whichever occurs first. Soft tissue disease status was assessed at regular intervals during the course of the study by CT of chest and CT or MRI of abdomen and pelvis. Results as of 03 Oct 2022 are reported for this outcome measure.
Time Frame: From the start of treatment to the time of first documented progression, or death (maximum up to 38 months)
Population: Included DDR-deficient participants randomized to double-blind study treatment in Part 2 regardless of whether or not treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part 2 Participants With DDR Deficiencies: Talazoparib+Enzalutamide: Participants with DDR deficiencies were randomized to receive talazoparib 0.5 mg QD in combination with enzalutamide 160 mg QD (up to a maximum of 169.86 weeks for both talazoparib and enzalutamide as of 03 Oct 2022).
- Part 2 Participants With DDR Deficiencies: Placebo+Enzalutamide: Participants with DDR deficiencies were randomized to receive placebo QD in combination with enzalutamide 160 mg QD (up to a maximum of 157 weeks for both placebo and enzalutamide as of 03 Oct 2022).
Arm/Group | Part 2 Participants With DDR Deficiencies: Talazoparib+Enzalutamide | Part 2 Participants With DDR Deficiencies: Placebo+Enzalutamide
Number analyzed (Participants) | 200 | 199
Months | NA [21.9 to NA] — NA indicates not estimated due to less than half of participants meeting the criterion as of data cutoff date (03 Oct 2022). | 13.8 [11.0 to 16.7]
Statistical Analysis 1: Comparison: Part 2 Participants With DDR Deficiencies: Talazoparib+Enzalutamide vs Part 2 Participants With DDR Deficiencies: Placebo+Enzalutamide; The following statistical hypotheses was tested to address the primary objectives: H02: HRrPFS+ ≥1 vs H12: HRrPFS+ <1, where HRrPFS and HRrPFS+ are the hazard ratios (talazoparib in combination with enzalutamide vs. placebo in combination with enzalutamide) of rPFS based on BICR assessment in the DDR deficient population for Part 2 Cohort 2; Test type: Superiority; p < 0.0001, Log Rank — 1-sided; Hazard Ratio (HR) = 0.447, 95% CI 2-sided [0.328 to 0.610] — Hazard ratio was based on Cox proportional hazards model; under proportional hazards, hazard ratio < 1 indicates reduction in hazard rate in favor of Talazoparib+Enzalutamide compared to Placebo+Enzalutamide

ADVERSE EVENTS:
Time Frame: Post first dose of any study intervention through 28 days after the last dose of study intervention (up to a maximum of 236 weeks)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs. DDR-deficient participants included in both the analysis for Part 2 Cohorts 1 and 2 were counted in both cohorts.
Groups:
- Part 1: Talazoparib 1 mg QD+Enzalutamide: Participants initially received a starting dose of talazoparib 1 mg once daily (QD) in combination with enzalutamide 160 mg QD up until Day 66, then the dose of talazoparib was reduced to 0.5 mg QD based on results from a review of available safety and pharmacokinetic (PK) data (up to a maximum of 231.14 weeks for both talazoparib and enzalutamide as of 16 Aug 2022). All-cause mortality and adverse events are reported for participants who received at least 1 dose of study intervention.
- Part 1: Talazoparib 0.5 mg QD+Enzalutamide: Participants received talazoparib 0.5 mg QD in combination with enzalutamide 160 mg QD (up to a maximum of 180 weeks for talazoparib and 219.29 weeks for enzalutamide as of 16 Aug 2022). All-cause mortality and adverse events are reported for participants who received at least 1 dose of study intervention.
- Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer): Participants were randomized to receive talazoparib 0.5 mg QD in combination with enzalutamide 160 mg QD (up to a maximum of 186.14 weeks for both talazoparib and enzalutamide as of 16 Aug 2022). All-cause mortality are reported for participants who were randomly assigned to double-blind study treatment in Part 2 regardless of whether or not treatment was administered. Adverse events are reported for participants who received at least 1 dose of study treatment in Part 2 and was based on the actual treatment received.
- Part 2 Cohort 1: Placebo+Enzalutamide (All-comer): Participants were randomized to receive placebo QD in combination with enzalutamide 160 mg QD (up to a maximum of 182 weeks for both placebo and enzalutamide as of 16 Aug 2022). All-cause mortality are reported for participants who were randomly assigned to double-blind study treatment in Part 2 regardless of whether or not treatment was administered. Adverse events are reported for participants who received at least 1 dose of study treatment in Part 2 and was based on the actual treatment received.
- Part 2 Participants With DDR Deficiencies: Talazoparib+Enzalutamide: Participants with DDR deficiencies were randomized to receive talazoparib 0.5 mg QD in combination with enzalutamide 160 mg QD (up to a maximum of 169.86 weeks for both talazoparib and enzalutamide as of 03 Oct 2022). Participants who were DDR-deficient and received talazoparib+enzalutamide in Part 2 Cohort 1 were combined with participants enrolled in Part 2 Cohort 2 and included in the analysis for Part 2 Participants With DDR Deficiencies. All-cause mortality are reported for participants who were randomly assigned to double-blind study treatment in Part 2 regardless of whether or not treatment was administered. Adverse events are reported for participants who received at least 1 dose of study treatment in Part 2 and was based on the actual treatment received.
- Part 2 Participants With DDR Deficiencies: Placebo+Enzalutamide: Participants with DDR deficiencies were randomized to receive placebo QD in combination with enzalutamide 160 mg QD (up to a maximum of 157 weeks for both placebo and enzalutamide as of 03 Oct 2022). Participants who were DDR-deficient and received placebo+enzalutamide in Part 2 Cohort 1 were combined with participants enrolled in Part 2 Cohort 2 and included in the analysis for Part 2 Participants With DDR Deficiencies. All-cause mortality are reported for participants who were randomly assigned to double-blind study treatment in Part 2 regardless of whether or not treatment was administered. Adverse events are reported for participants who received at least 1 dose of study treatment in Part 2 and was based on the actual treatment received.
Arm/Group | Part 1: Talazoparib 1 mg QD+Enzalutamide | Part 1: Talazoparib 0.5 mg QD+Enzalutamide | Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer) | Part 2 Cohort 1: Placebo+Enzalutamide (All-comer) | Part 2 Participants With DDR Deficiencies: Talazoparib+Enzalutamide | Part 2 Participants With DDR Deficiencies: Placebo+Enzalutamide
All-Cause Mortality (participants affected / at risk) | 5/13 | 2/6 | 123/402 | 129/403 | 43/200 | 53/199
Serious Adverse Events (participants affected / at risk) | 6/13 | 3/6 | 157/398 | 107/401 | 60/198 | 40/199
Other Adverse Events (participants affected / at risk) | 13/13 | 6/6 | 377/398 | 351/401 | 190/198 | 182/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Talazoparib 1 mg QD+Enzalutamide (N=13) | Part 1: Talazoparib 0.5 mg QD+Enzalutamide (N=6) | Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer) (N=398) | Part 2 Cohort 1: Placebo+Enzalutamide (All-comer) (N=401) | Part 2 Participants With DDR Deficiencies: Talazoparib+Enzalutamide (N=198) | Part 2 Participants With DDR Deficiencies: Placebo+Enzalutamide (N=199)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 55 | 1 | 17 | 2
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 2 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1 | 2 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 4 | 1 | 1 | 1
Pneumonia necrotising (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 4 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 2 | 2 | 1
Aortic thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 5 | 2 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 3 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 1
Retinal exudates (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 4 | 5 | 0 | 2
Death (General disorders) | 0 | 0 | 3 | 3 | 0 | 1 — For SAEs as reported with the preferred term "death", these events refer to cases where the cause of death was reported as unknown per investigator.
Chest pain (General disorders) | 0 | 0 | 1 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 9 | 3 | 4 | 3
Sepsis (Infections and infestations) | 0 | 0 | 3 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 6 | 1 | 3 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 5 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 4 | 1 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 3 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood culture positive (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2 | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 3 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2 | 2 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 0 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 4 | 3 | 4 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 2 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Malignant spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 10 | 4 | 3 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2 | 5 | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 4 | 1 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Bladder stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bladder tamponade (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Urinary bladder rupture (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
COVID infection with complications (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 — Uncoded Term
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Talazoparib 1 mg QD+Enzalutamide (N=13) | Part 1: Talazoparib 0.5 mg QD+Enzalutamide (N=6) | Part 2 Cohort 1: Talazoparib+Enzalutamide (All-comer) (N=398) | Part 2 Cohort 1: Placebo+Enzalutamide (All-comer) (N=401) | Part 2 Participants With DDR Deficiencies: Talazoparib+Enzalutamide (N=198) | Part 2 Participants With DDR Deficiencies: Placebo+Enzalutamide (N=199)
Anaemia (Blood and lymphatic system disorders) | 10 | 4 | 258 | 70 | 127 | 30
Neutrophil count decreased (Investigations) | 8 | 0 | 142 | 28 | 64 | 13
Fatigue (General disorders) | 5 | 5 | 134 | 118 | 66 | 53
Platelet count decreased (Investigations) | 3 | 0 | 98 | 14 | 49 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 8 | 4 | 3 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 4 | 0 | 2
Bundle branch block right (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0
Eustachian tube disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 6 | 4 | 3 | 2
Extraocular muscle disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 2 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 7 | 2 | 81 | 50 | 40 | 34
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 57 | 55 | 24 | 22
Vomiting (Gastrointestinal disorders) | 5 | 1 | 28 | 22 | 15 | 10
Constipation (Gastrointestinal disorders) | 3 | 1 | 72 | 68 | 26 | 32
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 15 | 15 | 10 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 12 | 9 | 6 | 3
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 17 | 19 | 7 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 7 | 2 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 15 | 6 | 5 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Noninfective gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 3 | 1 | 0 | 1
Influenza like illness (General disorders) | 1 | 3 | 5 | 10 | 2 | 4
Non-cardiac chest pain (General disorders) | 1 | 0 | 12 | 11 | 4 | 5
Oedema peripheral (General disorders) | 0 | 1 | 42 | 24 | 14 | 12
Peripheral swelling (General disorders) | 0 | 1 | 4 | 6 | 3 | 3
Pyrexia (General disorders) | 2 | 0 | 28 | 12 | 18 | 4
Asthenia (General disorders) | 0 | 0 | 56 | 38 | 30 | 29
Malaise (General disorders) | 0 | 0 | 25 | 12 | 4 | 4
Hypersensitivity (Immune system disorders) | 1 | 0 | 3 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 3 | 4 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 18 | 10 | 10 | 10
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 2 | 4 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 18 | 11 | 6 | 1
Otitis media (Infections and infestations) | 1 | 0 | 1 | 3 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 2 | 10 | 5 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 5 | 3 | 4 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 22 | 19 | 8 | 11
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 2 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 6 | 6 | 4 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 3 | 68 | 58 | 24 | 24
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 6 | 3 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 2 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 30 | 15 | 12 | 4
Alanine aminotransferase increased (Investigations) | 1 | 0 | 12 | 19 | 9 | 5
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 11 | 21 | 6 | 5
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 6 | 13 | 4 | 5
Blood pressure increased (Investigations) | 1 | 0 | 0 | 2 | 2 | 2
Lymphocyte count decreased (Investigations) | 3 | 0 | 45 | 20 | 14 | 12
Serum ferritin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 40 | 33 | 18 | 17
Weight increased (Investigations) | 0 | 1 | 6 | 8 | 2 | 0
White blood cell count decreased (Investigations) | 6 | 0 | 88 | 18 | 37 | 15
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 23 | 8 | 12 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 16 | 12 | 13 | 8
Decreased appetite (Metabolism and nutrition disorders) | 7 | 3 | 86 | 63 | 40 | 28
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 7 | 5 | 2 | 3
Gout (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 7 | 11 | 5 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 20 | 21 | 12 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 17 | 7 | 4 | 4
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 58 | 79 | 25 | 44
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 87 | 71 | 39 | 43
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 25 | 24 | 10 | 13
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 8 | 3 | 2
Jaw disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 9 | 3 | 8 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 19 | 15 | 6 | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 24 | 24 | 9 | 13
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 11 | 13 | 5 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 35 | 34 | 10 | 15
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 2 | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 2 | 2 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4 | 1 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 6 | 4 | 2 | 3
Dizziness (Nervous system disorders) | 4 | 1 | 48 | 24 | 20 | 15
Dysarthria (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 26 | 15 | 17 | 7
Encephalopathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 0 | 36 | 37 | 12 | 22
Hypersomnia (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 8 | 7 | 7 | 3
Lethargy (Nervous system disorders) | 1 | 0 | 3 | 7 | 3 | 5
Memory impairment (Nervous system disorders) | 4 | 0 | 13 | 14 | 7 | 7
Neuralgia (Nervous system disorders) | 1 | 0 | 2 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 3 | 0 | 12 | 10 | 6 | 8
Presyncope (Nervous system disorders) | 1 | 0 | 6 | 3 | 2 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 2 | 7 | 1 | 2
Somnolence (Nervous system disorders) | 1 | 0 | 4 | 0 | 4 | 2
Spinal cord oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 7 | 3 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 3 | 5 | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 0 | 6 | 9 | 4 | 8
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 3 | 0 | 1
Depressed mood (Psychiatric disorders) | 1 | 1 | 2 | 4 | 5 | 2
Depression (Psychiatric disorders) | 2 | 0 | 15 | 9 | 5 | 7
Mood swings (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 6 | 1 | 2 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 4 | 4 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 29 | 24 | 16 | 13
Calculus bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 14 | 31 | 10 | 14
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 7 | 2 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 6 | 2 | 2 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 6 | 9 | 4 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 6 | 13 | 2 | 6
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 6 | 13 | 8 | 2
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 2 | 4 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 13 | 7 | 4 | 10
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 13 | 11 | 4 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 40 | 24 | 17 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 5 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 20 | 8 | 7 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 6 | 5 | 2 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 5 | 3 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 10 | 3 | 4 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 8 | 2 | 1 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0 | 1
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 33 | 10 | 14 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 13 | 9 | 6 | 5
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 15 | 12 | 3 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 0 | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 5 | 3 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 9 | 2 | 11
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 2 | 0 | 1 | 0
Embolism venous (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 0
Hot flush (Vascular disorders) | 2 | 1 | 47 | 54 | 23 | 28
Hypertension (Vascular disorders) | 1 | 0 | 55 | 61 | 36 | 38
Hypotension (Vascular disorders) | 2 | 0 | 10 | 4 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03395197/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT03395197/SAP_001.pdf